CLINICAL TRIAL: NCT02738645
Title: A Clinical Cohort Study of Pneumonia in Respiratory Intensive Care Unit
Status: Recruiting | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Xiao Tang, Dr, Beijing Chao Yang Hospital
Other Study IDs: Pneumonia RICU
Record Dates: First submitted 2016-03-26; First posted 2016-04-14 (Estimated); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pneumonia in RICU: The patients admit in RICU because of pneumonia.
  Interventions: Other: pneumonia

INTERVENTIONS:
Other: pneumonia

SUMMARY:
From 2003 when Severe Acute Respiratory Syndromes (SARS) appeared，many new types of respiratory viruses emerge in endlessly. Therefore, the epidemiology and the clinical character has changed quietly, especially severe pneumonia. This cohort study aim to obtain the contents of severe pneumonia patients in Respiratory Intensive Care Unit (RICU). Through the clinical data analysis, the investigators could get the information of the pneumonia caused by different reasons, such as morbidity and mortality, risk factors, clinical symptoms and radiographic changes, the respiratory support parameter and so on. The investigators hope the result could guide them do the clinical work of severe pneumonia better in the future.

ELIGIBILITY:
Inclusion Criteria:

* admit in RICU because of pneumonia of any causes
* anticipated length of hospital stay more than 72h

Exclusion Criteria:

* admit in RICU because of other causes except pneumonia
* do not agree to join this study
* admit in RICU for the second time
* anticipated length of hospital stay less than 72h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients of RICU
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-06; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the mortality caused by any reasons in RICU | one years
the morbidity caused by any reasons in RICU | one years

SECONDARY OUTCOMES:
the symptoms description of pneumonia caused by any reasons in RICU | the first 48hours after admitted in RICU
  all the symptoms caused by pneumonia, such as fever, cough, dyspnea, sputum and so on. The investigators could get the incidence of each of these symptoms.
the respiratory support of pneumonia caused by any reasons in RICU | the first 5 days after admitted in RICU
  summarize the respiratory support parameters while the patients hospitalized in RICU. For example, the ventilation parameter and mode, Whether the mechanical ventilation complications occurred, and so on.
the treatment options of pneumonia caused by any reasons in RICU | 3 weeks
  the investigators obtain the treatment commons, such as the kind of antibiotics, the dosage of glucocorticoids, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, Dr, Principal Investigator — Beijing Chao-Yang Hospital, China
Locations (1):
- Department of respiratory and critical care medicine,Beijing Chao-yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided